CLINICAL TRIAL: NCT03518814
Title: Evaluation of the Quality of Life in Patients With Multimetastatic Melanoma Currently in Remission
Brief Title: Quality of Life in Patients With Multimetastatic Melanoma Currently in Remission (QUALM)
Acronym: QUALM
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0062
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Melanoma (Skin) Stage IV; Remission
Keywords: Melanoma stage IV; Remission; Quality of life
MeSH Terms: conditions — Melanoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multimetastatic melanoma in remission: Questionnaires
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — FACT-M (Functional Assessment of Cancer Therapy - Melanoma) questionnaire, MOS SF (medical outcome study short form) -36 questionnaire

SUMMARY:
Few studies have been conducted on the quality of life of patients with stage IV melanoma. Particularly, there is no data regarding the quality of life of patients with a multimetastatic melanoma currently in remission.

Then, the main objective of this study is to evaluate the quality of life from a point of view medico-psycho-social in patients with multimetastatic melanoma in remission for more than 6 months.

DETAILED DESCRIPTION:
The cutaneous melanoma, (9th rank of all cancers), was until recently neglected and poorly known by the general public. The metastatic stages have dramatic rates of survival: 25% at 1 year and 2% at 5 years with a median of about 6.2 months. However, in the last ten years, the treatment of metastatic forms has undergone a real revolution.

Its high metastatic potential for a very low initial tumor mass, gives evidence of a great aggressiveness. The cutaneous melanoma is resistant to the main therapeutics (chemotherapy and radiotherapy). Thanks to the emergence of immunotherapies and targeted therapies anti-RAF (Rapidly Accelerated Fibrosarcoma) and anti-MEK (Mitogen-activated Extracellular) the prognosis of patients with metastatic melanoma has considerably improved, increasing the number of "long-term survivors".

However, these treatments can cause many adverse effects that can impact patients' quality of life, despite a better tolerance compared to conventional chemotherapies. To our knowledge there are no data regarding the quality of life of patients with metastatic melanoma currently in remission.For this purpose, it is necessary to obtain solid data using validated questionnaires. Thus, we have chosen to evaluate quality of life using specific questionnaires to better understand patients' expectations, their difficulties, and then to improve the relationship between the patient and the physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Presenting a stage IV melanoma of the American Joint Committee on Cancer (AJCC) classification (multimetastatic) in remission for more than 6 months:
* Complete remission (defined as the complete disappearance of target lesions according to the RECIST criteria, based on a thoraco-abdomino-pelvic CT scan and a brain Magnetic resonance imaging (MRI) or
* Complete metabolic remission (defined as the complete disappearance of target lesions in PET CT (positron emission tomography computed tomograph, that is to say, disappearance of the hypermetabolic character of the anatomic structures. There may remain target lesions in conventional CT but they are not hypermetabolic in PET CT)
* Patients able to answer the questionnaires
* Patients with enough understanding of the French language

Exclusion Criteria:

* Adjuvant treatment
* Patient under tutorship or curatorship
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multimetastatic melanoma currently in remission
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Quality of life assessed by the Functional Assessment of Cancer Therapy-Melanoma (FACT-M) questionnaire | day 0
  The FACT-M questionnaire is a specific quality of life scale for patients treated for melanoma. It includes 51 items grouped into nine multi-item scores: six subscale scores and three summary scores.
  The six subscales consist of four subscales from the FACT-G:
  * physical well-being [PWB], score range: 0-28, higher values represent a worse outcome.
  * social well-being [SWB], score range: 0-28, higher values represent a better outcome.
  * emotional well-being [EWB], score range: 0-24, higher values represent a worse outcome.
  * functional well-being [FWB]), score range: 0-28, higher values represent a better outcome.
  One Melanoma scale, score range: 0-64, higher values represent a worse outcome. One Melanoma surgery scale, score range: 0-32, higher values represent a worse outcome.
  The three summary scores include:
  * the FACT-M Trial Outcome Index (TOI), score range: 0-120
  * the FACT-G total score, score range: 0-108
  * the FACT-M total score, score range: 0-172
Health status surveyed by the Medical Outcome Study Short Form - 36 (MOS SF 36) questionnaire | day 0
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
  The eight sections are:
  * vitality
  * physical functioning
  * bodily pain
  * general health perceptions
  * physical role functioning
  * emotional role functioning
  * social role functioning
  * mental health

CONTACTS AND LOCATIONS:
Overall Officials: Aurore Le Guern, Principal Investigator — Lille Catholic University
Locations (2):
- France (2):
  - Lille Catholic Hospitals, Lille, Nord
  - CHRU Lille, Lille, Nord

IPD SHARING:
Plan to Share IPD: No